CLINICAL TRIAL: NCT02359253
Title: Robot-Aided Diagnosis, Passive-Active Arm Motor and Sensory Rehabilitation Post Stroke: Aims 2&3
Brief Title: Robot Aided Rehabilitation - Intervention
Acronym: Aim2&3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); North Carolina State University (Other)
Responsible Party: Principal Investigator, Li-Qun Zhang, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00076764
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; Spasticity; Arm; Hand; Robotic therapy
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Muscle Stretching Exercises; Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IntelliArm with passive stretching (Experimental): Groups are split into 2 conditions based on stretching and 2 conditions based on target of intervention (arm or hand). Subjects will complete up to 30 minutes of strong passive stretching, then followed by 45-60 minutes of active movement training with the IntelliArm.
  Interventions: Other: Passive stretching; Other: IntelliArm
- IntelliArm with passive movement (Experimental): Groups are split into 2 conditions based on stretching and 2 conditions based on target of intervention (arm or hand). Subjects will wear the IntelliArm for up to 30 minutes with gentle passive movement or little stretching, then followed by 45-60 minutes of active movement training with the IntelliArm.
  Interventions: Other: Passive movement; Other: IntelliArm
- The hand robot with passive stretching (Experimental): Groups are split into 2 conditions based on stretching and 2 conditions based on target of intervention (arm or hand). Subjects will complete up to 30 minutes of strong passive stretching, then followed by 45-60 minutes of active movement training with the hand robot.
  Interventions: Other: Passive stretching; Other: Hand robot
- The hand robot with passive movement (Experimental): Groups are split into 2 conditions based on stretching and 2 conditions based on target of intervention (arm or hand). Subjects will wear the hand robot for up to 30 minutes with gentle passive movement or little stretching, then followed by 45-60 minutes of active movement training with the hand robot.
  Interventions: Other: Passive movement; Other: Hand robot

INTERVENTIONS:
Other: Passive stretching — Prior to active training, subjects will be passively move their arm or hand by IntelliArm or the hand robot within preset ranges of motion.
  Arms: IntelliArm with passive stretching; The hand robot with passive stretching
Other: Passive movement — Prior to active training, subjects will be passively move their arm or hand by IntelliArm or the hand robot only within ranges that produce no to very minimal forces.
  Arms: IntelliArm with passive movement; The hand robot with passive movement
Other: IntelliArm — During the active training, subjects will be asked to actively move their arm while supported with IntelliArm robot to interact with virtual targets and objects. The IntelliArm may provide resistance or assistance.
  Arms: IntelliArm with passive movement; IntelliArm with passive stretching
Other: Hand robot — During the active training, subjects will be asked to actively open and close their hand with the hand robot on while participating in task oriented occupational therapy focused on grasp and release tasks. The hand robot may provide resistance or assistance.
  Arms: The hand robot with passive movement; The hand robot with passive stretching

SUMMARY:
Sensorimotor impairments following stroke often involve complex pathological changes across multiple joints and multiple degrees of freedom of the arm and hand, thereby rendering them difficult to diagnose and treat. The objective of this study is to evaluate multi-joint neuromechanical impairments in the arm and hand, then conduct impairment-specific treatment, and determine the effects of arm versus hand training and the effects of passive stretching before active movement training.

DETAILED DESCRIPTION:
Sensorimotor impairments following stroke can lead to substantial disability involving the upper extremity. These impairments often involve complex pathological changes across multiple joints and multiple degrees-of-freedom of the arm and hand, thereby rendering them difficult to diagnose and treat. Many potential mechanisms, such as weakness, motoneuronal hyperexcitability, and elevated passive impedance, can contribute and it is currently unclear where to focus treatment. The objectives of this study are to address allocation of therapy resources between the arm and hand and to examine the benefits of combining passive stretching with active movement training.

Aim 1. To compare the efficacy of training the arm versus the hand in promoting upper extremity rehabilitation.

Hypothesis 1: Treating the proximal larger joints in the arm alone will lead to greater improvement than treating the distal hand alone.

Aim 2. To examine the efficacy of combining passive stretching with active (assistive or resistive) training for the shoulder, elbow, wrist, and hand.

Hypothesis 2: Multi-joint intelligent stretching followed by active (assistive or resistive) movement facilitated by use of the IntelliArm arm rehabilitation robot and a Hand rehabilitation robot will improve motor control of the upper extremity more than standard movement therapy alone.

Subjects will be assigned randomly with equal chance to one of four groups. Groups are split into 2 conditions based on stretching and 2 conditions based on target of intervention (arm or hand). Half of all the subjects will be assigned to the stretching groups and the other half to the passive movement groups. Half of the subjects will be assigned to the arm-training and the remaining half to hand-training groups. Arm-training groups will use the IntelliArm, hand-training groups will use the hand robot. For those assigned to the stretching groups, subjects will complete up to 30 minutes of passive stretching with the IntelliArm or the hand robot. For those assigned to the passive movement condition, subjects will do the robot according to their group assignment and wear it for up to 30 minutes with little to no stretching preceding the active therapy session. For each group, the initial about 30 minutes of stretching or relaxing will be followed by 45-60 minutes of active therapy with the IntelliArm or hand robot (depending on group assignment), for a total session time of 75-90 minutes.

The 4 groups of subjects will be compared against each other.

ELIGIBILITY:
Inclusion Criteria:

* First focal unilateral lesion, ischemic or hemorrhagic
* Had a stroke 1-12 months prior to enrollment
* Rated between stages 2-4 on the Chedoke McMaster Stroke Assessment Impairment Inventory: Stage of Recovery of the Arm and Hand

Exclusion Criteria:

* Apraxia
* Score of less than 22 on the Mini Mental Status Exam
* Severe pain in the shoulder by a self-rating of 7 out of 10 or greater
* Severe contracture in the upper extremity
* Unable to sit in a chair for 3 consecutive hours
* Unrelated musculoskeletal injuries
* Poor fit into equipment used in study
* Botox injection in upper extremity within 4 months
* Concurrent participation in gait or upper extremity intervention studies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-10-14 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline Graded Wolf Motor Function Test (WMFT) at two time points | Within 2 week prior to intervention, 2 week following intervention, and 2 months following intervention
  The WMFT is a quantitative measure of upper extremity motor ability through timed and functional tasks.

SECONDARY OUTCOMES:
Changes from baseline Fugl-Meyer Upper Extremity at two time points | Within 2 week prior to intervention, 2 week following intervention, and 2 months following intervention
  The Fugl-Meyer Assessment is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
Changes from baseline Chedoke McMaster Stroke Assessment: Impairment Inventory of Arm and Hand at two time points | Within 2 weeks prior to intervention, 2 weeks following intervention, and 2 months following intervention
  The Chedoke-McMaster Stroke Assessment (CMSA) is a screening and assessment tool utilized to measure physical impairment and activity of an individual following a stroke. The Chedoke Arm and Hand Activity Inventory (CAHAI) is used to assess functional ability of the paretic arm and hand. Each domain is scored on a 7-point scale.
Changes from baseline Modified Ashworth Scale (MAS) at two time points | Within 2 weeks prior to intervention, 2 weeks following intervention, and 2 months following intervention
  The Modified Ashworth Scale is the most widely used assessment tool to measure resistance to limb movement in a clinic setting. Scores range from 0-4, with 6 choices. 0 (0) - No increase in muscle tone; 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension; 1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM (range of movement); 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved; 3 (4) - Considerable increase in muscle tone passive, movement difficult; 4 (5) - Affected part(s) rigid in flexion or extension.
Changes from baseline Action Research Arm Test (ARAT) at two time points | Within 2 weeks prior to intervention, 2 weeks following intervention, and 2 months following intervention
  ARAT assesses the ability to handle objects differing in size, weight and shape and therefore can be considered to be an arm-specific measure of activity limitation.
Changes from baseline Grip Strength & Pinch Strength at two time points | Within 2 weeks prior to intervention, 2 weeks following intervention, and 2 months following intervention
  A dynamometer is used to measure grip strength and a pinch gauge to measure tip, key, and palmar pinch.
Changes from baseline Nottingham Sensory Assessment at two time points | Within 2 weeks prior to intervention, 2 weeks following intervention, and 2 months following intervention
  The assessment tests the tactile sensation of the patient through light touch, pressure and pinprick.
Changes from baseline range of motion (ROM) at two time points | Within 2 weeks prior to intervention, 2 weeks following intervention, and 2 months following intervention
  The range of motion (ROM) of shoulder, elbow, wrist and fingers will be measured in Degree.
Changes from baseline spasticity at two time points | Within 2 weeks prior to intervention, 2 weeks following intervention, and 2 months following intervention
  Spasticity will be measured by the resistance torque in Newton-meter under controlled movement at each joint.
Changes from baseline relaxation time of the finger flexor muscles at two time points | Within 2 weeks prior to intervention, 2 weeks following intervention, and 2 months following intervention
  Relaxation time will be quantified in Second by examining flexor muscle activity. The subject will be instructed to grip maximally upon hearing an audible tone. The subject should then relax his/her grip as quickly as possible after hearing a second tone. The relaxation time is defined as the elapsed time in Second from the second tone to the point at which the flexor muscle magnitude returns to the baseline level + three standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Qun Zhang, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):e6-e245. doi: 10.1161/CIR.0b013e31828124ad. Epub 2012 Dec 12. No abstract available. PMID 23239837
- [Background] Haggard P, Wing A. Coordinated responses following mechanical perturbation of the arm during prehension. Exp Brain Res. 1995;102(3):483-94. doi: 10.1007/BF00230652. PMID 7737394
- [Background] Hoffmann G, Schmit BD, Kahn JH, Kamper DG. Effect of sensory feedback from the proximal upper limb on voluntary isometric finger flexion and extension in hemiparetic stroke subjects. J Neurophysiol. 2011 Nov;106(5):2546-56. doi: 10.1152/jn.00522.2010. Epub 2011 Aug 10. PMID 21832028
- [Background] Kamper DG, Harvey RL, Suresh S, Rymer WZ. Relative contributions of neural mechanisms versus muscle mechanics in promoting finger extension deficits following stroke. Muscle Nerve. 2003 Sep;28(3):309-18. doi: 10.1002/mus.10443. PMID 12929190
- [Background] Kamper DG, Rymer WZ. Quantitative features of the stretch response of extrinsic finger muscles in hemiparetic stroke. Muscle Nerve. 2000 Jun;23(6):954-61. doi: 10.1002/(sici)1097-4598(200006)23:63.0.co;2-0. PMID 10842274
- [Background] Mayer NH, Esquenazi A, Childers MK. Common patterns of clinical motor dysfunction. Muscle Nerve Suppl. 1997;6:S21-35. PMID 9826981
- [Background] Shumway-Cook A, Woollacott MH (2001) Motor Control: Theory and Practical Applications, 2nd ed. vol. Chapter 6. Philadelphia: Lippincott Williams & Wilkins.
- [Background] Ren Y, Kang SH, Park HS, Wu YN, Zhang LQ. Developing a multi-joint upper limb exoskeleton robot for diagnosis, therapy, and outcome evaluation in neurorehabilitation. IEEE Trans Neural Syst Rehabil Eng. 2013 May;21(3):490-9. doi: 10.1109/TNSRE.2012.2225073. Epub 2012 Oct 19. PMID 23096119
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Gao F, Ren Y, Roth EJ, Harvey R, Zhang LQ. Effects of repeated ankle stretching on calf muscle-tendon and ankle biomechanical properties in stroke survivors. Clin Biomech (Bristol). 2011 Jun;26(5):516-22. doi: 10.1016/j.clinbiomech.2010.12.003. Epub 2011 Jan 6. PMID 21211873
- [Background] Wu YN, Hwang M, Ren Y, Gaebler-Spira D, Zhang LQ. Combined passive stretching and active movement rehabilitation of lower-limb impairments in children with cerebral palsy using a portable robot. Neurorehabil Neural Repair. 2011 May;25(4):378-85. doi: 10.1177/1545968310388666. Epub 2011 Feb 22. PMID 21343525
- [Background] Selles RW, Li X, Lin F, Chung SG, Roth EJ, Zhang LQ. Feedback-controlled and programmed stretching of the ankle plantarflexors and dorsiflexors in stroke: effects of a 4-week intervention program. Arch Phys Med Rehabil. 2005 Dec;86(12):2330-6. doi: 10.1016/j.apmr.2005.07.305. PMID 16344031
- [Background] Zhang LQ, Son J, Park HS, Kang SH, Lee Y, Ren Y. Changes of Shoulder, Elbow, and Wrist Stiffness Matrix Post Stroke. IEEE Trans Neural Syst Rehabil Eng. 2017 Jul;25(7):844-851. doi: 10.1109/TNSRE.2017.2707238. Epub 2017 May 23. PMID 28541901
- [Background] Zhang LQ, Xu D, Kang SH, Roth EJ, Ren Y. Multi-Joint Somatosensory Assessment in Patients Post Stroke. BMES Ann Meeting, Phoenix. 2017.